CLINICAL TRIAL: NCT03559933
Title: Percutaneous Electrical Phrenic Nerve Stimulation (PEPNS) System Feasibility Study
Brief Title: PEPNS System Feasibility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stimdia Medical Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIP0001
Record Dates: First submitted 2018-06-08; First posted 2018-06-18 (Actual); Results first posted 2021-09-16 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-07

CONDITIONS: Ventilator Induced Diaphragmatic Dysfunction (VIDD)

STUDY DESIGN:
Intervention Model Description: The pdSTIM Leads are temporarily inserted near the right and left phrenic nerves and connected to the PEPNS System console. Duration of stimulation in PEPNS study is up to 48 hours to allow periodic electrical stimulation in daily sessions until the patients is weaned or 48 hours since initiation of stimulation session has elapsed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- PEPNS System (Experimental): The pdSTIM lead will be temporarily inserted near the right and left phrenic nerves and connected to the PEPNS system console in order to stimulate the phrenic nerves and activate the diaphragm on the patients until extubated/removed from mechanical ventilation or until 48 hours has elapsed, whichever comes first.
  Interventions: Device: PEPNS System

INTERVENTIONS:
Device: PEPNS System — PEPNS System therapy will be delivered periodically up to 48 hours or less if patient is no longer being mechanically ventilated.
  Other Names: pdSTIM

SUMMARY:
The purpose of this feasibility study is to evaluate the safety and performance of the PEPNS System in patients that need to be mechanically ventilated for at least 48 hours and up to 7 days in the Intensive Care Unit (ICU).

DETAILED DESCRIPTION:
Mechanical ventilation is a life saving technology but can also cause damage to the lungs and diaphragm such as ventilator induced diaphragmatic dysfunction (VIDD). Research has shown that after being on mandatory mechanical ventilation and sedation the diaphragm begins to atrophy within as little as 18 hours. The PEPNS System consists of a console and disposable lead and will be used to stimulate the patient's diaphragm to contract in synchrony with the inspiratory cycle of the ventilator. The proprietary phrenic nerve to diaphragm stimulation (pdSTIM) Lead incorporates multipolar electrodes that align with the left and right phrenic nerves in order to stimulate the nerves to the diaphragm. This feasibility trial will investigate the safety and performance of the PEPNS System as a therapy by stimulating the diaphragm over a 48 hour period to facilitate weaning from the mechanical ventilator. The patient population includes those need to be mechanically ventilated for at least 48 hours and up to 7 days in the ICU.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years or older (Adult).
2. Able and willing to give informed consent or whose legally authorized representative is able and willing to give informed consent.
3. Subject who in the opinion of the admitting consultant/intensivist is likely to be ventilated for > 48 hours from time of recruitment since study treatment will be for up to 48 hours.

Exclusion Criteria:

1. Subject has a left ventricular ejection fraction (LVEF) < 20%.
2. Subject unlikely to survive 72 hours due to coexisting medical conditions.
3. Subject has an implanted pulse generator or implanted electronic device:
4. Subject has experienced an Acute Myocardial Infarction (AMI) within 72 hours prior to this screening or patient is on high dose inotropic support or subject is deemed to be in cardiogenic shock.
5. Subject has significant bleeding diathesis, or is at risk of significant haemorrhage, patient is receiving full dose systemic anticoagulation
6. Subject has a known or suspected phrenic nerve paralysis or neuromuscular or inflammatory muscle diseases where the diaphragm itself may not be functional.
7. Subject has an active systemic infection or local infection at or around the insertion site. Subject is neutropenic or has signs of significant immunocompromise.
8. Subject is known or suspected to be pregnant or is lactating.
9. Subject will be unavailable for, or is unwilling to comply with, follow up requirements of the protocol.
10. Subject is currently enrolled or is expected to be enrolled in any other study of an investigational drug or device who has received treatment under that protocol with the investigational product during the 30 days prior to screening.
11. Subject has undergone a surgery or interventional procedure within the neck region aside from placement of an internal jugular (IJ) vein catheter.
12. Subject has been diagnosed and has been treated for neck cancer within the past 5 years.
13. Subject is known to have a demonstrated intra cardiac thrombus on echocardiography.
14. Subject has uncontrolled hyperthyroidism, hypertension.
15. Subject has had any cerebral ischemic event (Stroke or Transient Ischemic Attack TIA) in the 6-month interval preceding the screening date.
16. Subject has degenerative nerve disorders such as amyotrophic laterals sclerosis (ALS).
17. Subject has an elevated hemidiaphragm on chest x-ray.
18. Subject written informed consent not obtained.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-07-10 (Actual); Primary Completion 2019-05-29 (Actual); Study Completion 2019-05-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michal M Soták, MD, Principal Investigator — Military University Hospital (UVN) Prague; James O'Rourke, PhD, Principal Investigator — Beaumont Hospital Dublin, Ireland
Locations (2):
- Military University Hospital (ÚVN), Prague, Czechia
- Beaumont Hospital, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: No
There will be no patient identifying information on any of the study case reports forms and all patients will only be identified by a study number.

REFERENCES:
- [Result] O'Rourke J, Sotak M, Curley GF, Doolan A, Henlin T, Mullins G, Tyll T, Omlie W, Ranieri MV. Initial Assessment of the Percutaneous Electrical Phrenic Nerve Stimulation System in Patients on Mechanical Ventilation. Crit Care Med. 2020 May;48(5):e362-e370. doi: 10.1097/CCM.0000000000004256. PMID 32191413
- [Derived] Sotak M, Roubik K, Henlin T, Tyll T. Phrenic nerve stimulation prevents diaphragm atrophy in patients with respiratory failure on mechanical ventilation. BMC Pulm Med. 2021 Oct 8;21(1):314. doi: 10.1186/s12890-021-01677-2. PMID 34625059
- See also: Initial Assessment of the Percutaneous Electrical Phrenic Nerve Stimulation System in Patients on Mechanical Ventilation — https://pubmed.ncbi.nlm.nih.gov/32191413/

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment Group: Percutaneous Electrical Phrenic Nerve Stimulation (PEPNS) Therapy: Stimdia Medical's pdSTIM L4300 leads will be inserted to lie close to the phrenic nerve in the neck region using ultrasound guidance into every patient who satisfies the Inclusion/Exclusion criteria and is enrolled in the study. Percutaneous electrical phrenic nerve stimulation (PEPNS) therapy will be administered via the Stimdia Medical PEPNS Console for six 2-hour sessions at 8-hour intervals over 48 hours, or until the patient is weaned; whichever comes first.
Period: Overall Study
Arm/Group | Treatment Group: Percutaneous Electrical Phrenic Nerve Stimulation (PEPNS) Therapy
Started (Date of first treatment for first treated patient (P01).) | 12
Completed (Date of follow-up visit for last treated patient (P12).) | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment Group: Percutaneous Electrical Phrenic Nerve Stimulation (PEPNS) Therapy
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.9 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 11
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 12
BMI [Mean (Standard Deviation); unit: kg/m^2] | 29.1 (6.6)
Neck Circumference at the Cricoid Cartilage [Mean (Standard Deviation); unit: centimeter] | 44.6 (5.3)

OUTCOME MEASURES:

1. Primary Outcome: Percent Capture of Left and/or Right Phrenic Nerve
Description: Capture of the Left and/or Right Phrenic Nerve > 80% with an output parameter of < 10.5 volts. Capture was defined as diaphragmatic movement as a direct consequence of electrical phrenic nerve stimulation. Capture for this analysis was defined as synchrony of the stimulated breath with the output parameter <10.5 volts and Work of Breath between 0.2 and 2.0 Joules/L. Synchrony was achieved if the lag time between start of inspiration and start of stimulation was less than 88 ms. The proportion of successful capture was analyzed using a generalized linear mixed model accounting for subject and stimulation within subject as random effects, and the outcome of capture was yes/no based on whether the stimulation captures the diaphragm with multiple observations per subject.
Time Frame: Up to 48 hours
Population: 10 patients with bilateral lead placement (excluding the initial two patients with left-sided lead placement only)
Measure: Number; unit: percentage of phernic nerve capture
Units Other Than Participants: Stimulated Breaths
Arm/Group | Treatment Group: Percutaneous Electrical Phrenic Nerve Stimulation (PEPNS) Therapy
Number analyzed (Participants) | 10
Number analyzed (Stimulated Breaths) | 36059
percentage of phernic nerve capture | 96.56
Statistical Analysis 1: Comparison: Treatment Group: Percutaneous Electrical Phrenic Nerve Stimulation (PEPNS) Therapy; The proportion of successful capture was analyzed using a generalized linear mixed model accounting for subject and stimulation within subject as random effects with multiple observations per subject. The null hypothesis was tested comparing the lower bound of the 98.75% two-sided confidence interval for the estimated percent diaphragm capture rate to the performance goal of 80%. If the lower bound was greater than 80%, the null hypothesis was rejected, and the endpoint was considered met; Test type: Superiority; p = 0.0125, Mixed Models Analysis; Subject and stimulation within subject as random effects with multiple observations per subject was accounted for; Logistic regression model = 95, 95% CI 2-sided [93.15 to 96.66], Standard Error of Mean 0.0152

2. Primary Outcome: Percent of Breaths Within Work of Breathing Range
Description: Work of Breathing (WOB) kept between 0.2 and 2.0 joules/L for 80% of stimulated breaths. Outcome is measured as a percentage of stimulated breaths that had a WOB between 0.2 joules/L and 2 joules/L and the performance goal was 80%.
Time Frame: Up to 48 hours
Measure: Number (95% Confidence Interval); unit: percentage of stimulated breaths
Units Other Than Participants: Stimulated Breaths
Arm/Group | PEPNS System
Number analyzed (Participants) | 10
Number analyzed (Stimulated Breaths) | 36059
percentage of stimulated breaths | 96.77 [96.58 to 96.95]

3. Secondary Outcome: Safe and Successful Lead Placement
Description: The percentage of patients who receive safe and successful placement of the multipolar lead in the left and right phrenic nerve utilizing ultrasound guidance will be determined.
Time Frame: Up to 48 hours
Measure: Number; unit: percentage of patients
Arm/Group | PEPNS System
Number analyzed (Participants) | 10
percentage of patients | 100

4. Secondary Outcome: Phrenic Nerve Stimulation Effectiveness
Description: Phrenic nerve stimulation in synchrony with Mechanical Ventilation breaths will be measured to verify that is occurs with inspiration.
Time Frame: Up to 48 hours
Measure: Number; unit: percentage of patients
Arm/Group | Treatment Group: Percutaneous Electrical Phrenic Nerve Stimulation (PEPNS) Therapy
Number analyzed (Participants) | 10
percentage of patients | 100

5. Secondary Outcome: Serious Device/Procedure Related Adverse Events
Description: The percentage of patients who experience one or more serious device/procedure-related adverse events during the study will be reported.
Time Frame: Up to 48 hours
Measure: Number; unit: percentage of patients
Arm/Group | Treatment Group: Percutaneous Electrical Phrenic Nerve Stimulation (PEPNS) Therapy
Number analyzed (Participants) | 10
percentage of patients | 0

ADVERSE EVENTS:
Time Frame: Adverse event data was collected during the therapy period (48 hours) and additional 30-37 days until follow-up.
Arm/Group | Treatment Group: Percutaneous Electrical Phrenic Nerve Stimulation (PEPNS) Therapy
All-Cause Mortality (participants affected / at risk) | 4/12
Serious Adverse Events (participants affected / at risk) | 4/12
Other Adverse Events (participants affected / at risk) | 0/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Group: Percutaneous Electrical Phrenic Nerve Stimulation (PEPNS) Therapy (N=12)
Patient Death (Nervous system disorders) | 4 (4) — Initial medical condition of subject at admission, despite intense medical care lead to subject death. Death unrelated to participation in the trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2018-11-30): https://cdn.clinicaltrials.gov/large-docs/33/NCT03559933/Prot_000.pdf
  • Statistical Analysis Plan (2019-03-19): https://cdn.clinicaltrials.gov/large-docs/33/NCT03559933/SAP_001.pdf
  • Informed Consent Form (2018-11-30): https://cdn.clinicaltrials.gov/large-docs/33/NCT03559933/ICF_002.pdf